CLINICAL TRIAL: NCT07255170
Title: DEVELOPMENT OF "GLYCEMIC CONTROL BAR WITH BEANS AND TOMATO FOR DIABETIC EATING" (GLYCOBITE) SNACK BAR FORMULATIONS AS A HEALTHY SNACK FOR DIABETES MELLITUS PATIENTS
Brief Title: RED BEAN AND TOMATO SNACK BAR FORMULATIONS AS A HEALTHY SNACK FOR DIABETES MELLITUS PATIENTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ngudi Waluyo (Other)
Responsible Party: Principal Investigator, Ummu Muntamah, Principal investigator, University Ngudi Waluyo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NgudiWaluyoUniversity
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus
Keywords: Blood glucose, diabetes mellitus, HbA1c, red beans, tomatoes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study comprise 100 participants who were randomly allocated to two groups. The GlycoBite group, consisting of 50 participants consuming 40 grams of "GlycoBite" snack bars daily and the control group consumed two packs of commercial snack bars, each weighing 20 grams. The intervention was conducted for 3 weeks.
  Weekly monitoring and evaluations were carried out. Interviews were done as part of the monitoring and evaluation procedure to find out 1) how compliant the participants were with snack bar consumption, 2) whether their activity changed, and 3) whether they had any complaints while eating. In the beginning, all participants had comprehensive history taking and clinical evaluation. Blood specimens were obtained following a 12-hour fasting period to assess the subsequent parameters at baseline and after treatment to evaluate blood glucose levels and HbA1c levels
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Patients in the control group consumed two packs of commercial snack bars, each weighing 20 grams every day. The intervention was conducted for 3 weeks.
  Interventions: Combination Product: The GlycoBite snack bar formula created is to combine tomatoes and red beans in a ratio of 60% and 40% respectively. Participants consuming 40 grams of "GlycoBite" snack bars daily
- Intervention group (Experimental): Participants consuming 40 grams of "GlycoBite" snack bars daily for 3 weeks.
  Interventions: Combination Product: The GlycoBite snack bar formula created is to combine tomatoes and red beans in a ratio of 60% and 40% respectively. Participants consuming 40 grams of "GlycoBite" snack bars daily

INTERVENTIONS:
Combination Product: The GlycoBite snack bar formula created is to combine tomatoes and red beans in a ratio of 60% and 40% respectively. Participants consuming 40 grams of "GlycoBite" snack bars daily — Participants consuming 40 grams of "GlycoBite" snack bars daily for 3 weeks

SUMMARY:
The goal of this clinical trial is to develop a "GlycoBite" snack bar formulation combination of red beans and tomatoes, and to assess its acceptability, nutritional content, and effectiveness on blood glucose levels in diabetic patients. The main questions it aims to answer are:

1. Dose snack bar formulation combination of red beans and tomatoes as a potensial healthy snack for diabetic patients?
2. Does snack bar formulation combination of red beans and tomatoes improve glycemic control
3. Does snack bar formulation combination of red beans and tomatoes lower blood glucose

DETAILED DESCRIPTION:
Researchers will compare GlycoBite (red beans and tomato combine) snack bar to commercial snack bar to see if GlycoBite works to control blood glucose

Participants will:

1. Take 40 grams of GlycoBite or commercial snack bar every day for 3 weeks
2. Weekly fasting blood glucose monitoring and evaluations were carried out.
3. Monitoring glycemic control ( HbA1c Levels) before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 DM patients
2. No medication therapy modifications during the intervention; and 4) no

Exclusion Criteria:

1. Other extreme diets
2. Severe stress or acute infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-22 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | Before intervention and every weeks for 3weeks ( Before intervention, in the first, secon and third weeks)
HbA1c meassure | Before intervention and 3 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ummu Muntamah, PhD, Principal Investigator — Ngudi Waluyo University; Medina Sianturi, PhD, Study Chair — Stikes E;;isabeth Semarang
Locations (1):
- Semarang, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leh HE, Mohd Sopian M, Abu Bakar MH, Lee LK. The role of lycopene for the amelioration of glycaemic status and peripheral antioxidant capacity among the Type II diabetes mellitus patients: a case-control study. Ann Med. 2021 Dec;53(1):1059-1065. doi: 10.1080/07853890.2021.1943515. PMID 34180336
- [Background] Has IM, Vodnar DC, Bungau AF, Tarce AG, Tit DM, Teleky BE. Enhanced Elderberry Snack Bars: A Sensory, Nutritional, and Rheological Evaluation. Foods. 2023 Sep 23;12(19):3544. doi: 10.3390/foods12193544. PMID 37835197
- [Background] Dimopoulou M, Vareltzis P, Floros S, Androutsos O, Bargiota A, Gortzi O. Development of a Functional Acceptable Diabetic and Plant-Based Snack Bar Using Mushroom (Coprinus comatus) Powder. Foods. 2023 Jul 14;12(14):2702. doi: 10.3390/foods12142702. PMID 37509794
- [Background] Md Isa Z, Ismail NH, Mohd Tamil A, Jaafar MH, Ismail R, Mohamed Noor Khan NA, Mat Nasir N, Ab Razak NH, Zainol Abidin N, Yusof KH. Pattern of macronutrients intake among type-2 diabetes mellitus (T2DM) patients in Malaysia. BMC Nutr. 2023 Jan 30;9(1):21. doi: 10.1186/s40795-022-00648-y. PMID 36717873
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Sievenpiper JL, Chan CB, Dworatzek PD, Freeze C, Williams SL. Nutrition Therapy. Can J Diabetes. 2018 Apr;42 Suppl 1:S64-S79. doi: 10.1016/j.jcjd.2017.10.009. No abstract available. PMID 29650114
- [Background] Kabiruyunusa A, Abdullahi N, Aliyu A. Kinetics of the thermal degradation of lycopene in tomatoes. Croat J Food Sci Technol 2020;12:84-9. https://doi.org/10.17508/cjfst.2020.12.1.11.
- [Background] Zaddana C, Nurmala S, Oktaviyanti T. Snack Bar Berbahan Dasar Ubi Ungu dan Kacang Merah sebagai Alternatif Selingan untuk Penderita Diabetes Mellitus Snack Bar Based on Purple Sweet Potato and Red Bean as an Alternative Snack for Diabetes Mellitus. Amerta Nutr 2021;1:260-75. https://doi.org/10.20473/amnt.v5i3.2021.
- [Background] Capanoglu E, Beekwilder J, Boyacioglu D, De Vos RC, Hall RD. The effect of industrial food processing on potentially health-beneficial tomato antioxidants. Crit Rev Food Sci Nutr. 2010 Nov;50(10):919-30. doi: 10.1080/10408390903001503. PMID 21108072
- [Background] Li M, Wang B, Lv W, Lin R, Zhao D. Characterization of pre-gelatinized kidney bean (Phaseolus vulgaris L.) produced using microwave hot-air flow rolling drying technique. Lwt 2022;154:112673. https://doi.org/10.1016/j.lwt.2021.112673.
- [Background] Ali MY, Sina AA, Khandker SS, Neesa L, Tanvir EM, Kabir A, Khalil MI, Gan SH. Nutritional Composition and Bioactive Compounds in Tomatoes and Their Impact on Human Health and Disease: A Review. Foods. 2020 Dec 26;10(1):45. doi: 10.3390/foods10010045. PMID 33375293
- [Background] Sianturi M, Susilaningsih N, Nugroho H, Suryani M. Lycopene Improves the Metformin Effects on Blood Glucose and Neutrophil Counts in Type 2 Diabetic Rats. Indones J Med Lab Sci Technol 2023;5:80-9. https://doi.org/10.33086/ijmlst.v5i1.3865.
- [Background] Leh HE, Lee LK. Lycopene: A Potent Antioxidant for the Amelioration of Type II Diabetes Mellitus. Molecules. 2022 Apr 4;27(7):2335. doi: 10.3390/molecules27072335. PMID 35408734
- [Background] Khan UM, Sevindik M, Zarrabi A, Nami M, Ozdemir B, Kaplan DN, Selamoglu Z, Hasan M, Kumar M, Alshehri MM, Sharifi-Rad J. Lycopene: Food Sources, Biological Activities, and Human Health Benefits. Oxid Med Cell Longev. 2021 Nov 19;2021:2713511. doi: 10.1155/2021/2713511. eCollection 2021. PMID 34840666
- [Background] Zhang Y, Bai Z, Xi X, Yang K, Yue C, Li P, Zhang K, Gao H, Guo J, Luo D. Influence of long-chain inulin phosphate monoester on structural and antidiabetic characteristics of red kidney bean steamed bread. Int J Biol Macromol. 2025 May;308(Pt 3):141965. doi: 10.1016/j.ijbiomac.2025.141965. Epub 2025 Mar 17. PMID 40101828
- [Background] Xu S, Qin L, Mazhar M, Zhu Y. Functional components profile and glycemic index of kidney beans. Front Nutr. 2022 Nov 2;9:1044427. doi: 10.3389/fnut.2022.1044427. eCollection 2022. PMID 36407530
- [Background] Dimopoulou M, Bargiota A, Barmpa E, Outskouni Z, Stagos D, Trachana V, Androutsos O, Gortzi O. Postprandial Glucose Response in Type 2 Diabetes Mellitus Patients and Possible Antioxidant Properties of a Plant-Based Snack Bar. Foods. 2024 Dec 20;13(24):4123. doi: 10.3390/foods13244123. PMID 39767064
- [Background] Ramírez-Jiménez AK, Gaytán-Martínez M, Morales-Sánchez E, Loarca-Piña G. Functional properties and sensory value of snack bars added with common bean flour as a source of bioactive compounds. Lwt 2018;89:674-80. https://doi.org/10.1016/j.lwt.2017.11.043.
- [Background] Gbolagade O, Oluwajuyitan T, Aderinola T, Oyeleye S, Oboh G, Fagbemi TN. Quality assessment and in-vivo glycemic indices of snack bar from blends of plantain our, soy cake, and oat bran. Discov Food 2024. https://doi.org/10.1007/s44187-024-00200-w.
- [Background] Nidhi Chauhan, Payal Mahajan. Snack Bars as a Functional Snack Option for Individuals with Diabetes: A Review. Indian J Public Heal Res Dev 2024;15:218-22. https://doi.org/10.37506/28ct9r25.
- [Background] Alhalabi B, Joseph A, Venkatasubramanian P. Nutritional values of ready-to-eat snacks available in the Indian E-market-a comparative study based on the health star rating system. Discov Food 2024;4. https://doi.org/10.1007/s44187-024-00087-7.
- [Background] Ummu M, Puji P, Hardhono S, Annastasia E LD. A Qualitative Study of Perceptions and Experiences of Living with a Diagnosis of Diabetes Mellitus. J Ilmu Keperawatan Komunitas 2023;6:1-19.
- [Background] Quarta A, Guarino M, Tripodi R, Giannini C, Chiarelli F, Blasetti A. Diet and Glycemic Index in Children with Type 1 Diabetes. Nutrients. 2023 Aug 9;15(16):3507. doi: 10.3390/nu15163507. PMID 37630698
- [Background] Chen L, Liu B, Ren L, Du H, Fei C, Qian C, Li B, Zhang R, Liu H, Li Z, Ma Z. High-fiber diet ameliorates gut microbiota, serum metabolism and emotional mood in type 2 diabetes patients. Front Cell Infect Microbiol. 2023 Jan 30;13:1069954. doi: 10.3389/fcimb.2023.1069954. eCollection 2023. PMID 36794003
- [Background] Long BY, Liang X. Dietary management of gestational diabetes: A review. Medicine (Baltimore). 2024 Jul 12;103(28):e38715. doi: 10.1097/MD.0000000000038715. PMID 38996126
- [Background] He P, Li H, Ye Z, Liu M, Zhou C, Wu Q, Zhang Y, Yang S, Zhang Y, Qin X. Association of a Healthy Lifestyle, Life's Essential 8 Scores With Incident Macrovascular and Microvascular Disease Among Individuals With Type 2 Diabetes. J Am Heart Assoc. 2023 Sep 5;12(17):e029441. doi: 10.1161/JAHA.122.029441. Epub 2023 Aug 23. PMID 37609934
- [Background] Ambroz M, de Vries ST, Buitenhuis G, Frost J, Denig P. Willingness of people with type 2 diabetes to engage in healthy eating, physical activity and medication taking. Prim Care Diabetes. 2024 Jun;18(3):347-355. doi: 10.1016/j.pcd.2024.03.006. Epub 2024 Apr 4. PMID 38575398